CLINICAL TRIAL: NCT05240014
Title: Enhancing Voluntary Motion in Broad Patient Populations With Modular Powered Orthoses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Robert D Gregg, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00201957; R01EB031166 (NIH)
Record Dates: First submitted 2022-01-13; First posted 2022-02-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lower-limb Orthoses; Frailty/Sarcopenia; Chronic Overuse Musculoskeletal Injuries
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Exoskeleton (Experimental): Participants in this arm of the study will perform various tasks while wearing the modular powered orthosis
  Interventions: Device: Modular powered orthosis

INTERVENTIONS:
Device: Modular powered orthosis — This study will investigate modular, lower-limb, powered orthoses that fit to user-specific weakened joints and control force/torque in a manner that enhances voluntary motion in broad patient populations. The central hypothesis is that high-torque, low-inertia motor systems controlled with energetic objectives will enable modular powered orthoses to partially assist the joints. High-torque electric motors combined with minimal transmissions can be freely rotated (i.e., backdriven) by human joints, allowing the use of an emerging torque control method called energy shaping to reduce the perceived weight/inertia of the body during any motion. By mounting these modular actuators to commercial orthoses, this technology will be easily prescribed/configured by clinicians.

SUMMARY:
The overall goal of this project is to develop modular, lower-limb, powered orthoses that fit to user-specific weakened joints and control force/torque in a manner that enhances voluntary motion in broad patient populations. This project aims to establish feasibility of assisting different populations with these modular powered orthoses. The investigators hypothesize that assisting lower-limb musculature with modular powered orthoses will improve 1) lifting/lowering posture in able-bodied subjects and 2) functional outcomes in elderly subjects.

DETAILED DESCRIPTION:
The overall goal of this project is to develop modular, lower-limb, powered orthoses that fit to user-specific weakened joints and control force/torque in a manner that enhances voluntary motion in broad patient populations. Conventional orthoses tend to immobilize joints, and emerging powered orthoses constrain voluntary motion by using highly geared electric motors and/or control methods that force the user to follow a specific gait pattern. Consequently, these devices have not seen widespread success across populations with weakened voluntary control due to advanced age, musculoskeletal disorders, etc. These heterogeneous populations require partial, not full, assistance of user-specific muscle groups during daily activities. However, there is a fundamental gap in knowledge about how to design and control powered orthoses to assist the user without constraining their motion. The central hypothesis of this project is that high-torque, low-inertia motor systems controlled with energetic objectives will enable modular powered orthoses to partially assist the joints. High-torque electric motors combined with minimal transmissions can be freely rotated (i.e., backdriven) by human joints, allowing the use of an emerging torque control method called energy shaping to reduce the perceived weight/inertia of the body during any motion. By mounting these modular actuators to commercial orthoses, this technology will be easily prescribed/configured by clinicians. This project aims to establish feasibility of assisting different populations with modular powered orthoses. The investigators hypothesize that assisting lower-limb musculature with modular powered orthoses will improve 1) lifting/lowering posture in able-bodied subjects and 2) functional outcomes in elderly subjects.

ELIGIBILITY:
Inclusion criteria for able-bodied, young participants will be:

* Aged between 18 to 65 years
* Weigh less than 250 lbs due to limitations in the design of the orthoses
* Ability to lift and lower a 10 kg weight using the neutral-spine squat technique for 10 repetitions

Exclusion criteria for able-bodied, young adult participants will be:

* Pregnant (self-report)
* Any significant neuromuscular or musculoskeletal disorder that would interfere with the study
* Prior history of chronic lower-back pain
* Unable to walk for 20 minutes
* History of any cardiovascular, vestibular, or visual diseases and/or impairments that may interfere with the study
* Cognitive deficits that would impair their ability to give informed consent or impair their ability to follow simple instructions during the experiments. Cognitive deficits will be determined by a Mini-Mental State Examination (MMSE) score of <22.
* Adults with a known allergy to medical grade tape

Inclusion criteria for elderly participants will be:

* Aged between 65 to 85 years
* Weigh less than 250 lbs due to limitations in the design of the orthoses
* Ability to walk 6 minutes without assistance from a person (may use walking aid)

Exclusion criteria for elderly participants will be:

* Pregnant (self-report)
* Significant pain due to arthritis or other joint problems that would limit their ability to walk
* Any recent lower-extremity fracture (within 3 months)
* Significant neurological (e.g., stroke), orthopedic, or cardiovascular disorder that may affect the ability to walk
* Advised by a physician not to walk or exercise
* Uncontrolled hypertension or diabetes
* Cognitive deficits or visual impairment that would impair their ability to give informed consent or impair their ability to follow simple instructions during the experiments. Cognitive deficits will be determined by a Mini-Mental State Examination (MMSE) score of <22.
* Adults with a known allergy to medical grade tape

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Powered orthosis effect (muscle effort) | 1 day
  For each orthosis module tested, electromyography (EMG) readings will be normalized per-muscle by the peak EMG observed during the no-orthosis condition, and then averaged over the cycle and across repetitions to obtain "normalized exertion" values. Performance will be assessed by the difference between the orthosis condition and no-orthosis condition, averaging across tasks and muscles measured for the joint module.
Time to complete 10 reps of lifting/lowering | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  Time to complete 10 reps of L&L will be measured post-fatigue in healthy subjects.
Gait speed | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  Gait speed will be determined by the time to complete a 10-meter walk test. This will be the primary outcome measure for elderly subjects.
Powered orthosis effect (biological torque) | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  For each orthosis module tested, peak biological torque (estimated by inverse dynamics) will be averaged across repetitions. Performance will be assessed by the difference between the orthosis condition and no-orthosis condition, averaging across tasks.
Minimum chair height for successful sit-to-stand | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  We will evaluate the minimum chair height from which elderly participants can successfully rise with and without the knee exoskeleton.
Joint power | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  For elderly participants, we will evaluate the peak values of biological and total (exo+biological) joint power with and without the exoskeleton.

SECONDARY OUTCOMES:
User satisfaction | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  User satisfaction / perception of device effectiveness over an ambulation circuit (sit-to-stand, walk up and down a ramp, walk up and down a staircase) will be measured post-fatigue in healthy subjects using a modified Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) survey. The purpose of the scale is to evaluate user device satisfaction and consists of 12 items asking the user to rate their satisfaction on a scale of 1 to 5, where 1 = "not satisfied at all" and 5 = "very satisfied".
Thorax angle | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  This is the global thorax angle (with respect to vertical) during a lifting/lowering cycle. This will be a secondary outcome measure for able-bodied subjects.
Stair ascent gait style | 1 day, assessed per experimental condition (i.e. with orthosis and without orthosis)
  Step-to-step vs. step-over-step gait style will be evaluated for the exo condition vs no exo condition for elderly participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab Lab, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided